CLINICAL TRIAL: NCT07012330
Title: A Multicenter Phase II Randomized Controlled Trial Comparing 177Lu-Dotatate/Capecitabine Combination Treatment With 177Lu-Dotatate in Neuroendocrine Tumor Patients
Brief Title: Comparing 177Lu-Dotatate/Capecitabine Combination Treatment With 177Lu-Dotatate in Neuroendocrine Tumor Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the number of dropouts and slow recruitment
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Morticia N. Becx, Coordinating investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2005-266
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine (NE) Tumors
Keywords: neuroendocrine tumor; peptide receptor radionuclide therapy; capecitabine; RCT
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors | interventions — Capecitabine; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 177Lu-Dotatate and capecitabine (Experimental): Patients with advanced somatostatin receptor positive gastroenteropancreatic (GEP) neuroendocrine tumors (NET) or bronchopulmonary NET were included to receive four cycles of 7.4 GBq 177Lu-Dotatate and capecitabine (1650 mg/m2/day) was administered for two weeks from the start of each peptide receptor radionuclide therapy (PRRT) cycle.
  Interventions: Drug: Capecitabine (Xeloda); Drug: 177Lu-DOTATATE
- 177Lu-Dotatate (Active Comparator): Patients with advanced somatostatin receptor positive gastroenteropancreatic (GEP) neuroendocrine tumore (NET) or bronchopulmonary NET were included to receive four cycles of 7.4 GBq 177Lu-Dotatate.
  Interventions: Drug: 177Lu-DOTATATE

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — Capecitabine (1650 mg/m2/day) was administered for two weeks from the start of each PRRT cycle.
  Arms: 177Lu-Dotatate and capecitabine
Drug: 177Lu-DOTATATE — Patients with advanced somatostatin receptor positive GEP NET or bronchopulmonary NET were included to receive four cycles of 7.4 GBq 177Lu-Dotatate.

SUMMARY:
Peptide receptor radionuclide therapy (PRRT) with [177Lu]Lu-[DOTA0,Tyr3]octreotate (177Lu-Dotatate) is an effective and safe treatment for patients with metastatic gastroenteropancreatic neuroendocrine tumors (GEP NET). While 177Lu-Dotatate prolongs progression-free survival (PFS) and preserves quality of life (QoL), objective response rates (ORR) remain limited. Capecitabine, as radiosensitizer, could increase efficacy without increasing 177Lu-Dotatate activity. This phase II randomized controlled trial investigated the additional cytotoxic or radiosensitizing effect of capecitabine in combination with 177Lu-Dotatate.

Patients with advanced somatostatin receptor positive GEP NET or bronchopulmonary NET were included to receive four cycles of 7.4 GBq 177Lu-Dotatate and capecitabine or 177Lu-Dotatate alone. Capecitabine (1650 mg/m2/day) was administered for two weeks from the start of each PRRT cycle. Primary endpoints were ORR, PFS and median overall survival (OS). Secondary endpoints included biochemical response, adverse events and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of histology proven GEP tumor(s), including bronchial carcinoids.
2. Presence of somatostatin-receptors on the known tumor lesions demonstrated by OctreoScan® within 6 months of the first dose of radiolabelled octreotate/octreotide. The uptake on the octreoscan should be at least as high as normal liver uptake on planar imaging.
3. Life expectancy greater than 12 weeks
4. Serum creatinine ≤150 μmol/liter or 1.7 mg/dL, and a measured creatinine clearance (or measured GFR using plasma clearance methods, not gamma-camera based) of ≥50 mL/min.
5. Hemoglobin (Hgb) concentration ≥5.5 mmol/L (≥8.9 g/dL); WBC ≥ 2*109/L (2000/mm3); platelets ≥ 100*109/L (100*103/mm3).
6. Total bilirubin ≤3 x ULN.
7. Serum albumin > 30 g/L, or serum albumin ≤ 30 g/L but normal prothrombin time.
8. Karnofsky Performance Status ≥ 60.
9. Presence of at least 1 measurable site of disease.
10. Patient's written voluntary informed consent to participate in the study, obtained prior to enrollment into the study. The informed consent must be maintained in the investigator's study files.

Exclusion Criteria:

1. Possible surgery with curative intent.
2. Surgery, radiotherapy, chemotherapy, or other investigational therapy within 3 months of the start of therapy.
3. Patients with known brain metastases unless these metastases have been treated and stabilized for at least six months prior to study start. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to study start.
4. Uncontrolled congestive heart failure.
5. Any subject who is taking concomitant medications which decrease renal function (such as aminoglycoside antibiotics).
6. Any subject receiving therapy with somatostatin analogues, unless the dose has been stable for at least 3 months prior to the first cycle in this study and the disease status during these 3 months has been documented by SWOG criteria as described in this study.
7. Any subject receiving therapy with short-acting somatostatin analogues in whom these analogues cannot be interrupted for 12 hours before and 12 hours after the administration of the radiolabelled somatostatin analogues, or any subject receiving therapy with long-acting somatostatin analogues in whom these analogues cannot be interrupted for at least 6 weeks before the administration of the radiolabelled somatostatin analogues, unless the uptake on the Octreoscan during continued somatostatin analogue medication is at least as high as normal liver uptake on planar imaging.
8. In patients with unusual hematological parameters, including an increased MCV (>105 fL), and especially in those who had previous chemotherapy, the advice of a hematologist should be seeked, for adequate further work-up.
9. Subjects with another significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
10. Pregnancy.
11. Prior radiation therapy to more than 25% of the bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rates | from enrollment until 2 years after treatment
  Radiological assessment
Progression-free survival | from enrollment until 2 years after treatment
  Radiological assessment
Overall survival | from enrollment until 2 years after treatment

SECONDARY OUTCOMES:
Biochemical response | from enrollment until 2 years after treatment
  Chromogranin A and alkaline phosphatase in the blood
Adverse events | from enrollment until 2 years after treatment
  Incidence and severity of adverse events according to CTCAE v5.0
Quality of life, Questioner | from enrollment until 2 years after treatment
  EORTC QLQ-30